CLINICAL TRIAL: NCT04400162
Title: Augmentation of Depression Treatment by Gamified Network Retraining: Feasibility, Effect Size Estimates, and User Experience
Brief Title: Augmentation of Depression Treatment by Gamified Network Retraining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Christian Plewnia, MD, Doctor of Psychiatry and Psychotherapy, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 248/2019BO1
Record Dates: First submitted 2020-01-09; First posted 2020-05-22 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Depression Mild; Cognitive Impairment; Cognitive Dysfunction; Depressive Disorder; Depression
MeSH Terms: conditions — Cognitive Dysfunction; Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCT (standard) (Active Comparator): This arm consists of the CCT in a standard variant that provides the basic training experience without any added gaming elements.
  Interventions: Behavioral: Usability of the CCT; Behavioral: Changes in regards to the depressive disorder
- CCT (game) (Experimental): This arm consists of the same CCT as the standard version, however pre-defined gaming elements that are thought to increase usability as well as interest in the intervention have been added.
  Interventions: Behavioral: Usability of the CCT; Behavioral: Changes in regards to the depressive disorder

INTERVENTIONS:
Behavioral: Usability of the CCT — Evaluation of the usability of the provided training.
Behavioral: Changes in regards to the depressive disorder — Evaluation of depressive symptoms and whether they change in regards to the provided training.

SUMMARY:
Major depressive disorder (MDD) is a highly prevalent and debilitating mental disorder with a high lifetime prevalence of 16-20%. Particularly for people with low socio-economic status, the existing and effective treatment options are hard to reach and show weaker effectivities. There is a potential to ameliorate depressive symptoms and improve quality of life in persons with mild-to-moderate depression by providing access to stimulating computerized trainings. Single computerized trainings that target depressive symptoms have been tested in laboratory and clinical settings so far. To date, innovative market access and confirmatory studies are missing for a large-scale implementation of such trainings. Thereby, the present work will foster a digitalized training paradigm (Paced-Auditory Serial Addition Task; PASAT) which was previously shown to reduce depressive symptoms, but in a novel innovative and gamified form on a tablet-PC handed out to participants. Different versions of the same training paradigm that comprise additional game elements will be compared. The feasibility study will gather data on effect size estimates of symptom severity reduction, user experience and usage in an ecological valid setting.

ELIGIBILITY:
Inclusion Criteria:

* Full age (> 18 years old)
* Consent
* German mother tongue
* Presence of mild-to-moderate depressive symptoms (MADRS > 10 and < 34 and confirmation of depressive symptoms in M.I.N.I. diagnostic interview)
* Stable or no medication with antidepressant drugs or other psychoactive agents (at least for 6 weeks)
* No or current psychotherapy

Exclusion Criteria:

* Presence of schizophrenia / psychotic disorder (according to M.I.N.I. diagnostic interview)
* Cognitive impairment
* Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Usability and feasibility on the UsExQ [User Experience Questionnaire] | 2-4 weeks
  Usage frequency, performed calculations during each session and over the course of the participation. Feedback on perceived quality of the device and software. Acceptance of training and willingness to continue (open text questionnaires; usability ranging from -- to ++ on a 5 point scale with negative responses corresponding to a more negative user experience).
MADRS [Montgomery-Asberg Depression Rating Scale] | 18-20 weeks
  Evaluation of depressive symptoms over the course of the intervention on the MADRS (lower numberes show decrease in depressive symptoms; range from 0-60).

SECONDARY OUTCOMES:
WHO-5 [WHO-Five Well-Being Index] (overall wellbeing) | 18-20 weeks
  Changes of the score over the course of the experiment (lower numbers showing decrease of perceived wellbeing; range from 0-25).
IDS-SR [Inventory of Depressive Symptomatology - Self Report] (depression) | 18-20 weeks
  Changes of the score over the course of the experiment (lower numbers showing decrease of symptoms; range from 0-84).
RSES [Rosenberg Self Esteem Scale] (self esteem) | 18-20 weeks
  Changes of the score over the course of the experiment (higher scores showing increase of self-esteem; range from 0-30).
SRQ [State Rumination Questionnaire] (rumination) | 18-20 weeks
  Changes of the score over the course of the experiment (lower scores showing decrease of ruminating thoughts; range from 10-50).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Plewnia, MD, Principal Investigator — University Hospital Tübingen
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weller S, Schroeder PA, Plewnia C. Gamification improves antidepressant effects of cognitive control training-A pilot trial. Front Digit Health. 2022 Oct 21;4:994484. doi: 10.3389/fdgth.2022.994484. eCollection 2022. PMID 36339520